CLINICAL TRIAL: NCT05900284
Title: A Randomized Clinical Trial of the Safety and Feasibility of Metformin as a Treatment for Sepsis Induced AKI.
Brief Title: Safety and Feasibility of Metformin for Sepsis Induced AKI
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Hernando Gomez (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Hernando Gomez, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY22120032; 1R01DK133142-01A1 (NIH)
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury; Metformin
Keywords: Sepsis; Septic Shock; Acute Kidney Injury; Metformin
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: One 500mg or 1,000mg tablet will be administered twice a day for the first (5) days of study treatment. One inactive tablet will be administered twice a day for the first (5) days of study treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties are blinded by participant group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin 500 mg (Experimental): One 500mg tablet will be administered twice a day for the first (5) days of study treatment.
  Interventions: Drug: Metformin low dose
- Placebo (Placebo Comparator): One inactive tablet will be administered twice a day for the first (5) days of study treatment.
  Interventions: Drug: Placebo
- Metformin 1,000 mg (Experimental): One 1,000mg tablet will be administered twice a day for the first (5) days of study treatment.
  Interventions: Drug: Metformin high dose

INTERVENTIONS:
Drug: Metformin low dose — If randomized to the 500 mg. Metformin arm, a tablet will be administered orally to the study participant twice a day for the initial five days starting on the date of study enrollment. Clinical research coordinators will collect blood and urine samples from study participants in both treatment arms. The blood will be collected at Baseline, Day 1 thru 7, and at hospital discharge or Day 30, whichever occurs first. On Day 2 and Day 5, the blood will be collected at hour-based intervals of 0.5h, 1h, 2h, 4h, 8h, 12h for a pharmacokinetic profile and delivered to the University of Pittsburgh Medical Center Clinical Laboratory for analysis. The remaining blood collection tubes will be delivered to the Clinical Research Biospecimen Core laboratory to be processed, separated into microtubes, and stored at -80°. Urine samples will be collected at Baseline, Day 1, 3, and 5. The urine will be processed, separated into microtubes, and frozen at -80°.
  Other Names: Glumetza low dose
  Arms: Metformin 500 mg
Drug: Metformin high dose — If randomized to the 1000 mg. Metformin arm, a tablet will be administered orally to the study participant twice a day for the initial five days starting on the date of study enrollment. Clinical research coordinators will collect blood and urine samples from study participants in both treatment arms. The blood will be collected at Baseline, Day 1 thru 7, and at hospital discharge or Day 30, whichever occurs first. On Day 2 and Day 5, the blood will be collected at hour-based intervals of 0.5h, 1h, 2h, 4h, 8h, 12h for a pharmacokinetic profile and delivered to the University of Pittsburgh Medical Center Clinical Laboratory for analysis. The remaining blood collection tubes will be delivered to the Clinical Research Biospecimen Core laboratory to be processed, separated into microtubes, and stored at -80°. Urine samples will be collected at Baseline, Day 1, 3, and 5. The urine will be processed, separated into microtubes, and frozen at -80°.
  Other Names: Glutzema high dose
  Arms: Metformin 1,000 mg
Drug: Placebo — If randomized to the Placebo arm, a tablet will be administered orally to the study participant twice a day for the initial five days starting on the date of study enrollment. Clinical research coordinators will collect blood and urine samples from study participants in both treatment arms. The blood will be collected at Baseline, Day 1 thru 7, and at hospital discharge or Day 30, whichever occurs first. On Day 2 and Day 5, the blood will be collected at hour-based intervals of 0.5h, 1h, 2h, 4h, 8h, 12h for a pharmacokinetic profile and delivered to the University of Pittsburgh Medical Center Clinical Laboratory for analysis. The remaining blood collection tubes will be delivered to the Clinical Research Biospecimen Core laboratory to be processed, separated into microtubes, and stored at -80°. Urine samples will be collected at Baseline, Day 1, 3, and 5. The urine will be processed, separated into microtubes, and frozen at -80°.
  Other Names: Placebo dose
  Arms: Placebo

SUMMARY:
Acute kidney injury (AKI) is an independent risk factor for death that affects 10-15% of hospitalized patients and more than 50% of patients admitted to the intensive care unit. Sepsis is the most frequent cause of AKI, affecting 48 million people worldwide every year, and accounting for approximately 11 million of annual global deaths. Despite these figures, there are no known therapies to prevent or reverse septic AKI; hence this study aims to establish the safety and feasibility of the implementation of metformin in the treatment of AKI in patients with sepsis.

This study is the first critical step to inform the design of a future, full-scale efficacy randomized clinical trial.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an independent risk factor for death, that affects 10-15% of hospitalized patients and more than 50% of patients admitted to the intensive care unit. The most frequent cause of AKI is Sepsis which affects 48 million people worldwide every year. Importantly, the 6-8-fold increase in the risk of death that AKI carries in sepsis, may be reversible because patients with sepsis who recover from AKI have similar 1- and 3-year mortality as those without AKI. These data agree with evidence showing that the development of AKI carries far-reaching consequences like remote organ dysfunction and an increased susceptibility to infection. These data suggest that AKI may be in the causal pathway to death from sepsis and that efforts to reverse AKI may improve the survival in patients with sepsis. However, there are no specific therapies to reverse or prevent the development of AKI during sepsis. Investigators have recently demonstrated that AMP-activated protein kinase (AMPK), a ubiquitous master regulator of cell metabolism and energy balance, is critical to protect the kidney from injury and enhance survival during experimental sepsis. Investigators have shown that pharmacologic activation of AMPK protects from AKI and improves survival, while inhibition increases kidney injury and death. Interestingly, metformin, the recommended first-line agent for the treatment of type 2 diabetes mellitus is a known AMPK activator. Based on this, investigators have demonstrated that treatment with metformin decreases mortality during experimental sepsis. Multiple observational human studies also support this idea. Two recent meta-analyses concluded that exposure to metformin was associated with a decreased risk of mortality. Investigators conducted the largest propensity-score matched retrospective study to date and demonstrated that metformin is associated with a decrease in the odds of moderate-severe AKI and death at 90-days, as well as with an increased odds of recovery from AKI. Despite this evidence, several gaps in knowledge remain. First, it is unclear if the protective effect of metformin is due to confounders. Second, it is unknown if the results of available studies are generalizable to non-diabetic patients.

Third, despite a track record of over 60 years of use in diabetic patients, safety has not been established in patients with septic shock. This proposal aims to conduct a randomized, placebo-controlled, feasibility study to establish the safety and feasibility of the use of oral metformin to prevent the development of sepsis-induced acute kidney injury and inform a future full-scale efficacy trial. Our overarching hypothesis is that in treatment of patients with sepsis, metformin is safe and effective in reducing sepsis-induced elevations in AKI biomarkers. Investigators will determine the safety of the use of metformin to treat adult patients with sepsis and will determine the pharmacokinetic profile of oral metformin (Aim 1), the feasibility of implementing this therapy (Aim 2) and estimate the heterogeneity of the effect of metformin on markers of kidney injury/stress and on circulating platelet mitochondrial function (Aim 3). This study is the first critical step to inform the design of a future, full-scale efficacy RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Admitted to the ICU with sepsis per sepsis 3 criteria (defined as suspected infection or initiation of anti-biotics plus an increase in SOFA ≥ 2 points)
3. Available enteral access

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2 prior to study drug administration
2. Not expected to survive more than 24 hours
3. Advanced directive to withhold life-sustaining treatment
4. Metformin use in the last 30 days from admission (assessed by medical or refill prescription history, and by medication reconciliation)
5. The treating clinician believes that participation in the trial would not be in the best interests of the patient
6. Known or suspected pregnancy
7. On mechanical circulatory support of any kind
8. History of allergy to metformin
9. Having severe metabolic acidosis defined by a venous or arterial pH < 7.2, with PaCO2 < 45 or PvCO2 < 50 mmHg at the time of enrolment.

   * Patients co-enrolled in observational studies will be eligible for enrollment in LiMiT AKI. However, patients enrolled in interventional studies will need to be assessed on an individual basis to define whether the patient will be eligible.
   * Children will be excluded from recruitment for this study. Etiologic causes of sepsis, acute kidney injury, and prognostic factors for children differ from those for adults; and for these reasons the proposed study focuses only on the adult population (age 18 years or older).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The development of metformin associated serious adverse events (mSAE) which will include hyperlactatemia, hypoglycemia, metabolic acidosis and/or gastrointestinal intolerance during the treatment period | Hospital discharge or 30 days, whatever occurs first
  Safety will be measured by monitoring the patient for the development of metformin associated serious adverse events (mSAE) which will include hyperlactatemia, hypoglycemia, metabolic acidosis and/or gastrointestinal intolerance during the treatment period. In addition, patients will be monitored for any adverse event or any significant adverse event.
Feasibility: Recruitment, retention and adherence | Hospital discharge or 30 days, whatever occurs first
  Investigators will quantify the number of patients screened and consented, the number of patients completing the study treatment, and the number of protocol deviations.
Feasibility: Investigating the reasons for denial of enrollment by patients, surrogates or clinicians | Hospital discharge or 30 days, whatever occurs first
  Investigators will identify barriers to implementing the intervention perceived by physicians, patients, or patients' surrogates who decline to participate or who drop out by requesting their feedback.
Feasibility: Data accrual and loss to follow-up | Hospital discharge or 30 days, whatever occurs first
  Investigators will estimate the proportion of randomized patients that achieve complete acquisition of outcome and ancillary data and lost to follow-up, and the proportion of missing data per variable.

SECONDARY OUTCOMES:
Area under the curve of the concentration of the renal biomarker TIMP2 (Time Point 2)/ Insulin-like growth factor-binding protein (IGFBP7) in time | Baseline, Day 1, 3, 5 to define the area under the concentration curve
  Investigators will measure the area under the curve of concentration of the tubular biomarker TIMP2/IGFBP7 vs. time using levels at baseline, day 1, 3 and 5.
Pharmacokinetic Accumulation Profile | Day 5
  Metformin accumulation levels will be assessed from study blood samples day 5 blood obtained at 0.5h, 1h, 2h, 4h, 8h, 12h, after administration of the last dose of Metformin.
Pharmacokinetic Absorption Profile | Day 2
  Metformin absorption kinetics will be assessed from study blood samples on Day 2, blood will be obtained at 0.5h, 1h, 2h, 4h, 8h, 12h, after first dose administration of Metformin.
Change in Platelet Mitochondrial Respiration | Change from baseline, Day 1, 3, 5
  Platelet bioenergetic profile will be assessed by measuring the oxygen consumption rate in the presence of sequential blockade of the different components of the electron transport chain using the SeaHorse analyzer on a subset of participants from each treatment arm.
Change in Platelet Mitochondrial Electron Transport Chain Complex Expression | Change from baseline, Day 1, 3, 5
  Platelet mitochondrial transport chain complex expression will be quantified by western blot using a LI-COR machine normalized to the Integrin alfa-2b protein.
Acute Kidney Injury at day 7 | At day 7
  AKI will be measured using the worse creatinine and urine output daily for 7 days and at discharge or day 30, whichever comes first.
Acute Kidney Injury at day 30 or discharge | Hospital discharge or day 30, whichever comes first.
  AKI will be measured using the worse creatinine and urine output daily for 7 days and at discharge or day 30, whichever comes first.
Number of patients requiring Renal Replacement Therapy within the hospitalization | Hospital discharge or 30 days, whichever comes first.
  Participants will be assessed on the need for any form of intermittent or continuous renal replacement therapy.
In-hospital Mortality | Hospital discharge or Day 30
  The proportion of patients who died while in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hernando Gomez, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The LiMiT-AKI study investigators will review the request for data from other investigators. The investigators will execute a data-sharing agreement with the University of Pittsburgh to share de-identified data with other investigators for research purposes only. The data sharing agreement will (ensure: i) a commitment to using the data only for research purposes and not to identify any individual data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After final enrolled participant is completed. Data will be shared for up to 12 months after the study is closed.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Saraiva IE, Hamahata N, Huang DT, Kane-Gill SL, Rivosecchi RM, Shiva S, Nolin TD, Chen X, Minturn J, Chang CH, Li X, Kellum J, Gomez H. Metformin for sepsis-associated AKI: a protocol for the Randomized Clinical Trial of the Safety and FeasibiLity of Metformin as a Treatment for sepsis-associated AKI (LiMiT AKI). BMJ Open. 2024 Apr 30;14(4):e081120. doi: 10.1136/bmjopen-2023-081120. PMID 38688665
- See also: BMJ Open Full Published Article — https://doi.org/10.1136/bmjopen-2023-081120